CLINICAL TRIAL: NCT07253077
Title: Evaluation of Cardiac and Endothelial Function Measured by Laboratory Biomarkers and Echocardiographic and Endothelial Testing in Children and Adolescents Treated With Anthracyclines
Brief Title: Evaluation of Cardiac and Endothelial Function in Children and Adolescents Treated With Anthracycline
Acronym: CARDIO-PED
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7304
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Anthracycline Related Cardiotoxicity in Childhood Cancers; Chemotherapeutic Toxicity; Childhood Cancer Survivors
Keywords: Childhood cancer survivors; Anthracycline related cardiotoxicity; Chemotherapy long term side effects; Cancer survivor follow up

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Peripheral blood samples for the measurement of biomarkers Serpin 3, THBS1, TGFbeta1, HIF1a, extracellular ICAM1, and endothelin
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated with anthracyclines: Patients who recovered from cancers and who underwent treatment with anthracyclines (from January 2010 to November 2024) and are undergoing regular follow-up. Inclusion criteria for the patient group:
  * diagnosis of hematologic oncology during childhood (diagnosis made between 0 and 16 years of age);
  * age at enrollment greater than or equal to 6 years;
  * having received anthracycline chemotherapy;
  * disease remission for at least 1 year;
  * absence of known cardiac disease prior to anthracycline therapy;
  * absence of congenital heart disease.
  Interventions: Diagnostic Test: Biomarker detection
- Control group: Subjects never treated with anthracyclines and free of cancer. Inclusion criteria for the control group:
  * Age at enrollment greater than or equal to 6 years;
  * Good health.
  Interventions: Diagnostic Test: Biomarker detection

INTERVENTIONS:
Diagnostic Test: Biomarker detection — All patients will be tested for plasma levels of Serpin 3, THBS1, TGFbeta1, HIF1a, extracellular ICAM1, and endothelin.
  In addition, the study will collect the following anamnestic data:
  * patient demographics, clinical data (age, sex, presence of comorbidities, medical history), instrumental data (echocardiogram performed), and laboratory data;
  * data relating to the neoplastic pathology and treatment performed
  Groups: Patients treated with anthracyclines
Diagnostic Test: Biomarker detection — All controls will be tested for plasma levels of Serpin 3, THBS1, TGFbeta1, HIF1a, extracellular ICAM1, and endothelin.
  In addition, the study will collect information on demographics, clinical data (age, sex, presence of comorbidities, medical history), instrumental data (echocardiogram performed), and laboratory data.
  Groups: Control group

SUMMARY:
In recent decades, the survival rate of children with cancer has increased significantly thanks to personalized treatments and the adoption of international therapeutic protocols. However, along with this increase in survival, side effects related to these treatments on various organs and systems have been observed.

Among the most widely used chemotherapeutic agents in pediatric age, anthracyclines play a crucial role in the treatment of various forms of neoplasms (both haematological such as acute lymphoblastic leukemia or lymphomas, and solid tumors such as sarcomas). However, in addition to their excellent antineoplastic effect, they are burdened by the potential for cardiotoxicity. This cardiotoxicity manifests clinically with left ventricular systolic dysfunction and arrhythmias.

At the moment, international guidelines recommend long-term cardiac follow-up evaluations for this group of patients, even after treatment has concluded.The methods used in the cardiac follow-up of patients undergoing anthracycline therapy include echocardiography, cardiac magnetic resonance imaging, tests to assess endothelial function, and measurements of the biomarkers troponin and atrial natriuretic peptide. These methods can assess anthracycline-induced cardiac and endothelial damage once it has already occurred, but they cannot predict its onset nor can they study its pathogenesis.

Furthermore, to date, no information is available regarding the possibility of using "endothelial-mesenchymal transition" biomarkers as predictors of the onset of anthracycline-induced cardiac damage.

This study analyzes these biomarkers as predictive tools for cardiac damage. Specifically, plasma levels of Serpin 3, THBS1, TGFbeta1, HIF1a, extracellular ICAM1, troponin, proBNP, fibrinogen, von Willebrand factor, and endothelin will be measured in patients treated with anthracycline. The concentrations of these biomarkers will be compared with the results of the echocardiogram and with the treatments performed in order to identify any relationships. Furthermore, plasma levels of Serpin 3, THBS1, TGFbeta1, HIF1a, extracellular ICAM1, troponin, proBNP, fibrinogen, von Willebrand factor, and endothelin will also be measured in a population of healthy subjects in order to obtain data on a possible relationship between the biomarkers and the anthracycline therapies performed.

ELIGIBILITY:
Inclusion Criteria for the patient group:

* diagnosis of cancer during childhood (diagnosis made between 0 and 16 years of age);
* age at enrollment greater than or equal to 6 years;
* having received anthracycline chemotherapy;
* disease remission for at least 1 year;
* absence of known cardiac disease prior to anthracycline therapy;
* absence of congenital heart disease.

Exclusion Criteria for the patient group:

* disease remission for less than 1 year;
* age less than 6 years at the time of enrollment;
* presence of known comorbidities (cardiopulmonary diseases, neurological diseases, etc.).

Inclusion Criteria for the control group:

* age at the time of enrollment: 6 years or older;
* good health.

Exclusion Criteria for the control group:

* having had oncological diseases;
* having undergone thoracic radiotherapy;
* having undergone anthracycline chemotherapy;
* being under 6 years of age at the time of enrollment;
* having known comorbidities (cardiopulmonary diseases, neurological diseases, etc.).

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The patient group will be selected among patients who have undergone anthracycline therapy and are undergoing regular follow-up at the Pediatric Oncology Unit of the Fondazione Policlinico Universitario A. Gemelli in Rome. Information about the tumor, treatments, and cardiac monitoring (echocardiogram) must be available for all patients. The control group will be selected from patients who visit the Pediatric Oncology Unit for a hematological evaluation but who have never undergone anthracycline therapy and have no known cardiac problems. All subjects (patients and controls) will undergo a thorough medical history and a clinical assessment, including a physical examination and measurement of vital signs and anthropometric parameters. Furthermore, all enrolled subjects, both patients and controls, will be required to collect, at a routine blood sampling time, a 6 ml tube for the measurement of biomarkers of endothelial-mesenchymal transition and endothelial activation.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To assess the possible presence of differences in the concentration of early biomarkers of "endothelial-mesenchymal transition" and endothelial damage between subjects treated with anthracycline therapy and healthy controls. | Biomarker assays will be performed only upon enrollment.
  Measurement of the concentration of biomarkers of endothelial-mesenchymal transition and endothelial damage (Serpin 3, THBS1, TGF-beta1, HIF1a, extracellular ICAM1, troponin, proBNP, fibrinogen, von Willebrand factor, endothelin) in patients who had recovered from cancer and underwent anthracycline therapy and compared with controls.
To evaluate possible associations between measured biomarkers and echocardiogram results and medical history in subjects treated with anthracycline therapy. | Biomarkers and medical history will be collected at the moment of enrollement in the study
  Measurement of the linear correlation between biomarkers and the results obtained in the echocardiographic examination and the treatments performed.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Ruggiero, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No